CLINICAL TRIAL: NCT06317324
Title: A Prospective, Single Center, Observational Study:Compare the Prognostic Differences Between SBRT and Surgery for NSCLC Patients With Interlobular Fissure Invasion.
Brief Title: Compare the Prognostic Differences Between SBRT and Surgery for NSCLC Patients With Interlobular Fissure Invasion.
Status: Recruiting | Type: Observational
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: bc2023200
Record Dates: First submitted 2024-03-10; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: NSCLC; Radiotherapy; Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgery Group: Diagnosed as primary lung cancer by imaging/pathology, meeting the indications for surgical treatment; The clinical staging is cIB-IIIB stage (cT2-3N0M0), regardless of whether the staging is overestimated or underestimated as confirmed by pathology.
- SBRT Group: Diagnosed as primary lung cancer by imaging/pathology, meeting the indications for SBRT treatment; The clinical staging is cIB-IIIB stage (cT2-3N0M0), regardless of whether the staging is overestimated or underestimated as confirmed by pathology.
  Interventions: Other: Different treatments

INTERVENTIONS:
Other: Different treatments — NSCLC patients receive the treatment of SBRT
  Groups: SBRT Group

SUMMARY:
The goal of this observational study is to compare the prognostic differences between SBRT and Surgery for NSCLC patients with interlobular fissure invasion. The main questions it aims to answer are:

1. Explore the survival differences.
2. Explore of the lung function changes before and after different treatments.

DETAILED DESCRIPTION:
Main purpose:

Explore the survival differences between SBRT and surgery for NSCLC patients with interlobular pleural invasion.

Secondary purpose:

1. Longitudinal exploration of the differences in heart and lung function changes before and after treatment between SBRT and surgery of NSCLC patients with interlobular pleural invasion
2. Longitudinal exploration of dynamic changes in lung lobe volume before and after treatment in NSCLC patients with interlobular pleural invasion treated with SBRT and surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate and sign an informed consent form in writing;
2. Age 18 and above, regardless of gender;
3. Diagnosed as primary lung cancer through imaging/pathology, meeting the indications for SBRT and surgical treatment;
4. The clinical staging is cIB-IIIB stage (cT2-3N0M0), regardless of whether the staging is overestimated or underestimated as confirmed by pathology;
5. Imaging diagnosis of NSCLC patients with tumor invasion of interlobular pleura;
6. No serious abnormalities in the blood system, heart, lungs, liver, kidney function, or immune deficiency;
7. There are no restrictions on surgical methods, and both VATS and open chest surgery are acceptable;
8. Physical condition score ECOG level 0-2;
9. Expected survival time>3 months.

Exclusion Criteria:

1. Pathological confirmation of small cell lung cancer;
2. Non solitary lung cancer, non primary lung cancer, with distant metastasis;
3. Individuals with a history of severe lung or heart disease;
4. Severe comorbidities, such as uncontrolled hypertension, heart failure, etc;
5. Pregnant or lactating women;
6. Previous history of malignant tumors;
7. Refusal or inability to sign the informed consent form for participating in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinically diagnosed cIB-IIIB stage (cT2-3N0M0) NSCLC patients and tumor invades Interlobular pleura.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
OS | 3 years
  Overall Survival
PFS | 3 years
  Progression Free Survival
MRFS | 3 years
  Distant Metatasis Free Survival
LRFS | 3 years
  Local Relapse Free Survival

SECONDARY OUTCOMES:
VC | 1 year
  Vital Capacity
FVC | 1 year
  Forced Vital Capacity
FEV1 | 1 year
  Forced Expiratory Volume in one second
DLCO | 1 year
  Diffusing Capacity of the lungs for carbon monoxide
PFR | 1 year
  Pulmonary Function Report

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin Key Laboratory of Cancer Prevention and Therapy, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided